CLINICAL TRIAL: NCT05589233
Title: Clinical Phenotype of Persons Vaccinated Against Sars-CoV-2 Hospitalized for COVID-19 Disease as a Basis for Optimalization of National Vaccination Strategy and Post-exposure Prophylaxis
Brief Title: COVID-19 Vaccination AZV 2021-2023
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Renata Černá Pařízková, doctor, University Hospital Hradec Kralove
Other Study IDs: AZVCR_FNHK_9302
Record Dates: First submitted 2022-10-20; First posted 2022-10-21 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: COVID-19; Vaccination; Immunity; Respiratory Failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients COVID-19 positive admitted to the hospital: COVID-19-positive patients admitted eighter to the standard ward or intensive care unit who were vaccinated against SARS-Cov-2
  Interventions: Biological: Vaccionation eighter started or full course

INTERVENTIONS:
Biological: Vaccionation eighter started or full course — Vaccination against SARS-CoV-2 at any number of doses

SUMMARY:
The study is aimed at the clinical and laboratory characteristics of patients with completed vaccination against SARS-CoV-2 admitted to the hospital in the standard ward and intensive care unit due to the severe course of COVID-19.

DETAILED DESCRIPTION:
The high number of patients hospitalized for COVID-19 significantly affects the entire healthcare system, where 70-80% of the total number of patients are unvaccinated, however, approximately 20-30% of patients hospitalized for the disease COVID-19 have undergone vaccination. The investigators assume the existence of several phenotypes of infection even in vaccinated patients, which may differ both in the rate of antibody formation, the dynamics of indicators of persistent virus replication, and the intensity of a potentially self-destructive inflammatory reaction and activation of coagulation. Early identification of patients with completed vaccination who have a higher risk of a severe course of COVID or a demonstrable inadequate immune response will allow individualization of treatment. Finding out the risk characteristics of the patients is a question and the difference in the type of vaccine on the severity of the course of hospitalization and the clinical outcome of the patients can contribute to the optimization of the vaccination strategy of the population and to the early identification of risk groups of vaccinated persons from the point of view of the timely deployment of available post-exposure prophylaxis/treatment procedures.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* COVID-19 positiveness
* vaccination against SARS-CoV-2 (any number of doses)

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the standard ward or intensive care unit with COVID-19 positive test and any number of vaccination doses against SARS-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Patient phenotype | 1.1.2021 - 30.6.2023
  Clinical and laboratory characteristics of patients with completed vaccination against SARS-CoV-2 admitted to the hospital in the standard ward and intensive care unit due to the severe course of COVID-19.

SECONDARY OUTCOMES:
Vaccination status | 1.1.2021 - 30.6.2023
  Defining the clinical phenotype of patients with completed vaccination against SARS-CoV-2 that is associated with the highest risk of severe course of the disease and/or death.
Vaccine efectiveness | 1.1.2021 - 30.6.2023
  Assessment of the difference between the effectiveness of the vaccines used in relation to the need for admission of patients to intensive care unit and indicators of clinical outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia